CLINICAL TRIAL: NCT06501989
Title: A Pilot Study of Pharmacokinetically (PK) Dose Adjusted 5-Fluorouracil (5-FU) in Patients With Metastatic Colorectal Cancer
Brief Title: Study of 5-fluorouracil (5-FU) in Patients With Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator has left Inova
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INOVA-2024-27
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: 5-fluorouracil (5-FU); pharmacokinetic assay
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Each cycle of chemotherapy is 2 weeks long, so you will be receiving treatment on the study for a total of 8 weeks. You will also need additional imaging (CT scans) after you complete the first four cycles of chemotherapy, which brings your total time in the study to about 3 months including treatment and follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy with 5-FU/Leucovorin (LV) alone, with oxaliplatin or irinotecan or both (Experimental): Plasma specimens will be collected for the measurement of plasma 5-FU level from patients receiving 5-FU/LV alone, with oxaliplatin (mFOLFOX6) or irinotecan (FOLFIRI), or both (mFOLFOXIRI) chemotherapy. 5-FU doses will be modified based on the assay results.
  Interventions: Drug: Biweekly 5-FLUOROURACIL (5-FU); Drug: Biweekly Modified FOLFOX6; Drug: Biweekly FOLFIRI; Drug: mFOLFOXIRI

INTERVENTIONS:
Drug: Biweekly 5-FLUOROURACIL (5-FU) — 5-FU 2400 mg/m². Infusion for 46 hours. Leucovorin 200 mg/m². Either a vascular endothelial growth factor (VEGF) inhibitor or epidermal growth factor (EGFR) inhibitor or may be added to the regimen at the discretion of the treating physician. Repeat every 2 weeks.
  Other Names: 5-FU
Drug: Biweekly Modified FOLFOX6 — Oxaliplatin 85 mg/m². 5-FU 400 mg/m² on day 1 as bolus (OPTIONAL). 5-FU 2400 mg/m² Infusion for 46 hours. Leucovorin 200 mg/m2. Repeat every 2 weeks
  Other Names: fluorouracil, leucovorin, oxaliplatin combined
Drug: Biweekly FOLFIRI — Irinotecan 180 mg/m2. 5-FU 400 mg/m2 on day 1 as bolus (OPTIONAL). 5-FU 2400 mg/m2 Infusion for 46 hours. Leucovorin 200 mg/m2.
  Repeat every 2 weeks.
  Other Names: irinotecan with fluorouracil (5FU) and folinic acid combined
Drug: mFOLFOXIRI — Irinotecan 165 mg/m2. Oxaliplatin 85 mg/m2. 5-FU 2400 mg/m2 Infusion for 46 hours. Repeat every 2 weeks.
  Other Names: folinic acid, fluorouracil (5FU), oxaliplatin, irinotecan combined

SUMMARY:
The purpose of this research is to see if adjusting the dose of 5-fluorouracil based on its concentration in your blood will improve the treatment of your metastatic colon cancer.

DETAILED DESCRIPTION:
5-fluorouracil (5-FU) has been the most widely used agent in the treatment of early stage and advanced colorectal cancer. Traditionally, 5-FU dosing is based on body surface area (BSA). However, BSA-dosing has been associated with a wide range of pharmacokinetic (PK) variability, resulting in marked differences in drug exposure and toxicities in an individual. There is a significant association between the risk of 5-FU-related toxicities and the extent of 5- FU systemic exposure, which can be measured using a well-established pharmacokinetic (PK) assay.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age.
* Histologically confirmed metastatic colorectal cancer eligible for treatment with 5-FU.
* No prior therapy for metastatic disease. If adjuvant 5-FU or FOLFOX was administered, the last dose must have been at least 6 months prior to the diagnosis of metastatic disease.
* Adequate organ function.
* Eastern Cooperative Oncology Group (ECOG) status less than or equal to 2.
* Life expectancy > 3 months.

Exclusion Criteria:

* Untreated brain metastasis. Treated brain metastases are allowed as long as symptoms have resolved off of steroids.
* At least 4 weeks from any prior surgery or 2 weeks from radiation treatments.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-19 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Feasibility Of Pharmacokinetically (PK) Guided Does Adjustment of 5-Fluorouracil (5-FU) In a Community Oncology Setting | From enrollment to the end of treatment at 8 weeks
  The Feasibility Of Pharmacokinetically Guided Does Adjustment of 5-Fluorouracil In a Community Oncology Setting is Defined as 80% Success Rate among Patients Who Has Completed Four Sequential PK blood Draws with Subsequent Dose Adjustments During the Treatment with 5-FU based Drug Therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Huynh, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Health Care Service, Falls Church, Virginia, United States

REFERENCES:
- [Background] Tournigand C, Andre T, Achille E, Lledo G, Flesh M, Mery-Mignard D, Quinaux E, Couteau C, Buyse M, Ganem G, Landi B, Colin P, Louvet C, de Gramont A. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004 Jan 15;22(2):229-37. doi: 10.1200/JCO.2004.05.113. Epub 2003 Dec 2. PMID 14657227
- [Background] Cremolini C, Antoniotti C, Rossini D, Lonardi S, Loupakis F, Pietrantonio F, Bordonaro R, Latiano TP, Tamburini E, Santini D, Passardi A, Marmorino F, Grande R, Aprile G, Zaniboni A, Murgioni S, Granetto C, Buonadonna A, Moretto R, Corallo S, Cordio S, Antonuzzo L, Tomasello G, Masi G, Ronzoni M, Di Donato S, Carlomagno C, Clavarezza M, Ritorto G, Mambrini A, Roselli M, Cupini S, Mammoliti S, Fenocchio E, Corgna E, Zagonel V, Fontanini G, Ugolini C, Boni L, Falcone A; GONO Foundation Investigators. Upfront FOLFOXIRI plus bevacizumab and reintroduction after progression versus mFOLFOX6 plus bevacizumab followed by FOLFIRI plus bevacizumab in the treatment of patients with metastatic colorectal cancer (TRIBE2): a multicentre, open-label, phase 3, randomised, controlled trial. Lancet Oncol. 2020 Apr;21(4):497-507. doi: 10.1016/S1470-2045(19)30862-9. Epub 2020 Mar 9. PMID 32164906
- [Background] Fang L, Xin W, Ding H, Zhang Y, Zhong L, Luo H, Li J, Yang Y, Huang P. Pharmacokinetically guided algorithm of 5-fluorouracil dosing, a reliable strategy of precision chemotherapy for solid tumors: a meta-analysis. Sci Rep. 2016 May 27;6:25913. doi: 10.1038/srep25913. PMID 27229175
- [Background] Meyerhardt JA, Mayer RJ. Systemic therapy for colorectal cancer. N Engl J Med. 2005 Feb 3;352(5):476-87. doi: 10.1056/NEJMra040958. No abstract available. PMID 15689586
- [Background] Gamelin E, Delva R, Jacob J, Merrouche Y, Raoul JL, Pezet D, Dorval E, Piot G, Morel A, Boisdron-Celle M. Individual fluorouracil dose adjustment based on pharmacokinetic follow-up compared with conventional dosage: results of a multicenter randomized trial of patients with metastatic colorectal cancer. J Clin Oncol. 2008 May 1;26(13):2099-105. doi: 10.1200/JCO.2007.13.3934. PMID 18445839
- [Background] Siegel RL, Miller KD, Fedewa SA, Ahnen DJ, Meester RGS, Barzi A, Jemal A. Colorectal cancer statistics, 2017. CA Cancer J Clin. 2017 May 6;67(3):177-193. doi: 10.3322/caac.21395. Epub 2017 Mar 1. PMID 28248415
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Background] Kaldate RR, Haregewoin A, Grier CE, Hamilton SA, McLeod HL. Modeling the 5-fluorouracil area under the curve versus dose relationship to develop a pharmacokinetic dosing algorithm for colorectal cancer patients receiving FOLFOX6. Oncologist. 2012;17(3):296-302. doi: 10.1634/theoncologist.2011-0357. Epub 2012 Mar 1. PMID 22382460
- [Background] Gamelin EC, Danquechin-Dorval EM, Dumesnil YF, Maillart PJ, Goudier MJ, Burtin PC, Delva RG, Lortholary AH, Gesta PH, Larra FG. Relationship between 5-fluorouracil (5-FU) dose intensity and therapeutic response in patients with advanced colorectal cancer receiving infusional therapy containing 5-FU. Cancer. 1996 Feb 1;77(3):441-51. doi: 10.1002/(SICI)1097-0142(19960201)77:33.0.CO;2-N. PMID 8630950
- [Background] Beumer JH, Boisdron-Celle M, Clarke W, Courtney JB, Egorin MJ, Gamelin E, Harney RL, Hammett-Stabler C, Lepp S, Li Y, Lundell GD, McMillin G, Milano G, Salamone SJ. Multicenter evaluation of a novel nanoparticle immunoassay for 5-fluorouracil on the Olympus AU400 analyzer. Ther Drug Monit. 2009 Dec;31(6):688-94. doi: 10.1519/JSC.0b013e3181b866d0. PMID 19935361
- [Background] Gamelin E, Boisdron-Celle M, Guerin-Meyer V, Delva R, Lortholary A, Genevieve F, Larra F, Ifrah N, Robert J. Correlation between uracil and dihydrouracil plasma ratio, fluorouracil (5-FU) pharmacokinetic parameters, and tolerance in patients with advanced colorectal cancer: A potential interest for predicting 5-FU toxicity and determining optimal 5-FU dosage. J Clin Oncol. 1999 Apr;17(4):1105. doi: 10.1200/JCO.1999.17.4.1105. PMID 10561167
- [Background] Morawska K, Goirand F, Marceau L, Devaux M, Cueff A, Bertaut A, Vincent J, Bengrine-Lefevre L, Ghiringhelli F, Schmitt A. 5-FU therapeutic drug monitoring as a valuable option to reduce toxicity in patients with gastrointestinal cancer. Oncotarget. 2018 Jan 30;9(14):11559-11571. doi: 10.18632/oncotarget.24338. eCollection 2018 Feb 20. PMID 29545919
- [Background] Wilhelm M, Mueller L, Miller MC, Link K, Holdenrieder S, Bertsch T, Kunzmann V, Stoetzer OJ, Suttmann I, Braess J, Birkmann J, Roessler M, Moritz B, Kraff S, Salamone SJ, Jaehde U. Prospective, Multicenter Study of 5-Fluorouracil Therapeutic Drug Monitoring in Metastatic Colorectal Cancer Treated in Routine Clinical Practice. Clin Colorectal Cancer. 2016 Dec;15(4):381-388. doi: 10.1016/j.clcc.2016.04.001. Epub 2016 May 7. PMID 27256667
- [Background] Kirkwood JM, Ensminger W, Rosowsky A, Papathanasopoulos N, Frei E 3rd. Comparison of pharmacokinetics of 5-fluorouracil and 5-fluorouracil with concurrent thymidine infusions in a Phase I trial. Cancer Res. 1980 Jan;40(1):107-13. PMID 7349890
- [Background] Au JL, Rustum YM, Ledesma EJ, Mittelman A, Creaven PJ. Clinical pharmacological studies of concurrent infusion of 5-fluorouracil and thymidine in treatment of colorectal carcinomas. Cancer Res. 1982 Jul;42(7):2930-7. PMID 6211226